CLINICAL TRIAL: NCT01978249
Title: A Randomized, Prospective, Multicenter Study for the Role of Primary Tumor Resection in Colorectal Cancer Patients With Asymptomatic, Synchronous Unresectable Metastasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the difficulties of participant enrollment.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0277
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Primary tumor resection; Chemotherapy; Overall survival; Quality of life
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy first without primary tumor resection (Experimental): Patients will receive chemotherapy first without primary tumor resection.
  Interventions: Procedure: Systemic chemotherapy
- Primary tumor resection followed by chemotherapy (Active Comparator): Patients will receive primary tumor resection followed by chemotherapy.
  Interventions: Procedure: primary tumor resection (PTR)

INTERVENTIONS:
Procedure: Systemic chemotherapy
  Arms: Chemotherapy first without primary tumor resection
Procedure: primary tumor resection (PTR) — primary tumor resection (PTR) using open or laparoscopy or robotic surgery
  Arms: Primary tumor resection followed by chemotherapy

SUMMARY:
Short description for lay public, include brief statement of the study hypothesis

ELIGIBILITY:
Inclusion Criteria:

* Age : between 20 and 90 years old
* Histologically confirmed adenocarcinoma of the colon or the upper rectum
* Patients with resectable primary colon or upper rectal cancer and unresectable metastatic lesions.
* Patients with no primary cancer related symptoms.
* ECOG performance status of 0 - 2
* Appropriate organ functions (hepatic transaminases - less than 5 times the normal range; bilirubin - less than 2 times the normal range; creatinine serum - less than 1.5 times the normal range; thrombocyte - more than 100,000/µl; neutrophil - more than 1,500/µl)
* ASA score of < 3
* An informed consent form has been signed by the patient.

Exclusion Criteria:

* The patient received adjuvant chemotherapy within the past 6 months.
* The patient received chemotherapy for metastatic colon cancer.
* The patient was planning to have curative surgery for the metastatic lesions.
* The primary cancer is unresectable.
* Patients with peritoneal carcinomatosis.
* Patients with mid and low rectal cancer (< 10cm)
* Patients with primary tumor related complications such as intestinal obstruction, intractable bleeding, and perforation, that needs to be treated.
* ASA score of > 4
* The patient has chronic hepatitis or cirrhosis. An asymptomatic HBV or HCV carrier can participate.
* Patients with an active infection, which need antibiotic therapy, during the randomization period.
* Pregnant or breastfeeding women
* Patients who were enrolled in another clinical trial during the time of enrollment (within the 28 day randomization period).
* Patients with another different malignant tumor during the past 5 years. Patients with treated non-melanoma skin cancer or cervical cancer can be enrolled in this study.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the overall survival between patients who underwent primary tumor resection and patients who received chemotherapy without primary tumor resection | 2 years after allocation
  Comparison of the overall survival between patients who underwent primary tumor resection followed by chemotherapy and patients who received chemotherapy without primary tumor resection in stage IV colorectal cancer patients with unresectable metastasis.

SECONDARY OUTCOMES:
Analysis of primary tumor related complications in the chemotherapy group and postoperative complications in the primary tumor resection followed by the chemotherapy group. | 2 years after allocation

OTHER OUTCOMES:
To compare the quality of life between the two groups using the Korean version of EORTC QLQ (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire)-C30. | 2 years after allocation

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - National Cancer Center, Ilsan, Gyeonggi-do
  - Gachon University, Gil Hospital, Incheon, Gyeonggi-do
  - Seoul National University, Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Yeongnam University Hospital, Daegu, Gyeongsang-do
  - Wonkwang University Hospital, Iksan, Jeollabukdo
  - Chonnam National University Hospital, Gwangju, Jeonlla Nam-do
  - Kyungpook National University Hospital, Daegu
  - Department of Surgery, Yonsei University College of Medicine, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University, Gangnam Severance Hospital, Seoul

REFERENCES:
- [Derived] Kim CW, Baek JH, Choi GS, Yu CS, Kang SB, Park WC, Lee BH, Kim HR, Oh JH, Kim JH, Jeong SY, Ahn JB, Baik SH. The role of primary tumor resection in colorectal cancer patients with asymptomatic, synchronous unresectable metastasis: Study protocol for a randomized controlled trial. Trials. 2016 Jan 19;17:34. doi: 10.1186/s13063-016-1164-0. PMID 26782254